CLINICAL TRIAL: NCT05783986
Title: Developing a MRI-based Deep Learning Model to Predict MMR Status of Endometrial Carcinoma
Brief Title: Developing a MRI-based Deep Learning Model to Predict MMR Status
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-084-01
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Endometrial Cancer
Keywords: deep learning, MMR, MRI
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Testing group: 375 patients of our hosipital,randomly divided.
  Interventions: Other: randomly divided
- Internal validation group: 125 patients of our hosipital,randomly divided.
  Interventions: Other: randomly divided
- External validation group: 100 patients of Sun Yat-sen University Cancer Center

INTERVENTIONS:
Other: randomly divided — 500 patients of our hospital were randomly divided into testing group and internal validation group, and 100 patients in collabrative hospital were external validation group.
  Groups: Internal validation group; Testing group

SUMMARY:
In order to develop a convenient, cheap and comprehensive method to preoperatively predict dMMR and reduce the number of people requiring dMMR-related immunohistochemical or genetic testing after surgery, this study aims to establish a deep learning model based on MRI to predict the MMR status of endometrial cancer. Patients diagnosed with endometrial cancer after surgery and who had completed pelvic MRI before surgery were collected. Deep learning was used to combine the clinical model with MR Image data to build the model. ROC curves were constructed for the testing group, internal verification group and external verification group, and the area under ROC curves were calculated to evaluate the diagnostic effect and stability of the model.

The dual threshold triage strategy was used to screen out the pMMR population (below the lower threshold), dMMR population (above the upper threshold) and the uncertain part of the population (between the thresholds).

DETAILED DESCRIPTION:
In this study, patients diagnosed with endometrial cancer after surgery and who had completed pelvic MRI before surgery were collected from 2017 to 2022. It is expected to collect 500 cases in our hospital, which are divided into 375 cases (experimental group) and 125 cases (internal verification group).

100 cases of Sun Yat-sen University Cancer Center for external verification. Clinical data (age, gender, BMI, CA125, CA19-9, MR-T staging, immunohistochemical results of MMR-related proteins) of the study population were collected and logistics regression analysis was conducted to establish clinical models. Extract, segment, integrate and enhance MR Image data.

Deep learning was used to combine the clinical model with MR Image data to build the model. ROC curves were constructed for the testing group, internal verification group and external verification group, and the area under ROC curves were calculated to evaluate the diagnostic effect and stability of the model.

The dual threshold triage strategy was used to screen out the pMMR population (below the lower threshold), dMMR population (above the upper threshold) and the uncertain part of the population (between the thresholds). If the predictive score is above the lower threshold, the patient is advised to undergo further immunohistochemical or genetic testing to confirm MMR status or dMMR type

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with endometrial cancer after surgery and who had completed pelvic MRI before surgery from 2017 to 2022

Exclusion Criteria:

* (1) There was no immunohistochemical detection result of MMR-related protein; (2) Radiotherapy and chemotherapy before MRI; (3) small tumors that are difficult to identify on the image (<5mm) ; (4) The T2-weighted imaging quality is insufficient to plot ROI, such as obvious motion artifacts; (5) There are other gynecological malignancies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with endometrial cancer after surgery and who had completed pelvic MRI before surgery
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-04-17 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under receiver operating characteristic curve (AUROC) | one year
  The area under receiver operating characteristic curve (AUROC) was used to evaluate the performance of the models

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No
there is not a plan to make individual participant data (IPD) available to other researchers.